CLINICAL TRIAL: NCT00132821
Title: Impact of Smoking Cessation on Sleep
Brief Title: Impact of Smoking Cessation on Sleep - 5
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: NIDA-16427-5; R01-16427-5; DPMC
Record Dates: First submitted 2005-08-18; First posted 2005-08-22 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2009-06

CONDITIONS: Tobacco Use Cessation; Sleep Disorders
Keywords: Nicotine dependence; Sleep disorders; smoking cessation; Relapse
MeSH Terms: conditions — Tobacco Use Cessation; Sleep Wake Disorders; Tobacco Use Disorder; Smoking Cessation; Recurrence | interventions — Bupropion; Tobacco Use Cessation Devices

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- A (Active Comparator): Bupropion
  Interventions: Drug: Bupropion
- B (Active Comparator): Transdermal nicotine patch
  Interventions: Drug: Transdermal Nicotine Patch
- C (Placebo Comparator)
  Interventions: Drug: Placebo Bupropion
- D (Placebo Comparator)
  Interventions: Drug: Placebo transdermal nicotine patch

INTERVENTIONS:
Drug: Bupropion — Days 1-3, 150 mg Bupropion in am; days 4-63, 300 mg Bupropion (150 mg in am and 150 mg in pm)
  Other Names: Zyban
  Arms: A
Drug: Transdermal Nicotine Patch — 21-mg nicotine patch applied in AM for 6 weeks, starting on the morning of quit day; 14-mg patch applied in AM for 2 weeks; 7-mg patch applied in AM for 1 week
  Arms: B
Drug: Placebo Bupropion — Days 1-3, 150 mg placebo Bupropion in am; days 4-63, 300 mg placebo Bupropion (150 mg in am and 150 mg in pm)
  Arms: C
Drug: Placebo transdermal nicotine patch — 21-mg placebo nicotine patch applied in AM for 6 weeks, starting on the morning of quit day; 14-mg placebo patch applied in AM for 2 weeks; 7-mg placebo patch applied in AM for 1 week
  Arms: D

SUMMARY:
Smoking is a major health problem with a direct link to elevated heart- and lung-related problems. Nicotine is highly addictive, which makes quitting difficult and relapse after quitting highly probable. Any type of sleep disturbance may make quitting even harder. The purpose of this study is to evaluate the effect of bupropion and nicotine replacement therapies (NRT) on sleep disturbances. In turn, this might show how such medications affect attempts at smoking cessation.

DETAILED DESCRIPTION:
The majority of attempts to quit smoking end in failure due to unpleasant withdrawal symptoms. One such symptom is sleep disturbances. Bupropion, effective in assisting with smoking cessation, commonly causes sleep disturbances as a medication side effect. In addition, a number of NRTs also cause sleep disturbances. This study will aim to characterize the effect of smoking cessation and smoking cessation treatments on sleep by measuring central and autonomic nervous system arousal. The study will also evaluate the impact of smoking cessation treatments on daytime sleepiness and mood as well as their effect on smoking relapse.

Participants will be randomly assigned to one of four groups. Participants will receive either bupropion (150 mg for 3 days and 300 mg for 60 days) or placebo, starting one week prior to smoking quit day. They will then receive either active NRT (21 mg for 6 weeks, 14 mg for 1 week, and 7 mg for 1 week) or placebo, starting on quit day. Participants will be studied for up to 5 nights in a sleep lab. Sleep studies will include polysomnography measurements, including electrooculography of both eyes, activity of mentalis muscle and both anterior tibialis muscles, EEG, ECG, oxygen saturation, airflow, and respiratory efforts. Sleep studies will occur on the 2 nights prior to quit day, the quit night, and the 2 nights after quitting. Each sleep study will be followed by daytime measures. These will include a series of self-report instruments, sleepiness and performance measures, and physiological activity measures. Carbon monoxide levels will also be a daytime measurement and must fall below 10 ppm on the post quit days. All participants will receive bimonthly phone counseling for 12 months, starting on quit day. Participants will have follow-up evaluations at Months 3 and 12 in order to measure carbon monoxide levels and complete self-report instruments.

ELIGIBILITY:
Inclusion Criteria:

* Meets DSM-IV criteria for nicotine dependence
* History of smoking at least 20 cigarettes each day for 2 years prior to enrollment
* Expired carbon monoxide level of at least 10 ppm
* Body mass index less than 30 kg/m2

Exclusion Criteria:

* Meets DSM-IV criteria for dependence on substances other than nicotine and caffeine
* Substance abuse within the year prior to enrollment
* History of DSM-IV diagnosis of schizophrenia, bipolar disorder, obsessive compulsive disorder, or chronic depression
* Current diagnosis of major depression
* History of neurological illness or trauma (e.g., stroke, seizure disorder, febrile seizures, electroconvulsive therapy)
* Family history of seizure disorder
* History of head injury with loss of consciousness for longer than 1 hour
* Currently diagnosed with a sleep disorder
* Currently diagnosed with anorexia or bulimia
* Severe or chronic cardiovascular, lung, kidney, or neurological disease
* Uncontrolled hypertension or diabetes
* Use of medications contraindicated with bupropion
* High frequency alcohol use or binge drinking in the month prior to enrollment
* Pregnant or breastfeeding

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2005-08; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Pre- and post-cessation sleep measures by in-laboratory polysomnography | Up to 7 days post-cessation

SECONDARY OUTCOMES:
Smoking cessation status confirmed by carbon monoxide levels | Up to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Gary Swan, Principal Investigator — SRI International
Locations (1):
- SRI International, Menlo Park, California, United States

REFERENCES:
- [Background] Colrain IM, Trinder J, Swan GE. The impact of smoking cessation on objective and subjective markers of sleep: review, synthesis, and recommendations. Nicotine Tob Res. 2004 Dec;6(6):913-25. doi: 10.1080/14622200412331324938. PMID 15801567